CLINICAL TRIAL: NCT04557306
Title: An Open, 3+3 Design With Dose De-escalation, Single-center, Phase 1 Trial to Evaluate Tolerabiility and Safety of Intravenously Administered CBT101, an Autologous Natural Killer Cell, in Patients Who Underwent Curative Surgery and Adjuvant Therapy for Solid Cancer
Brief Title: Evaluationn of Tolerability and Safety of CBT101, an Autologous Natural Killer Cell, in Patients With Solid Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CHABiotech CO., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CBT101_P1
Record Dates: First submitted 2020-09-15; First posted 2020-09-21 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-02

CONDITIONS: Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CBT101 q2w (Experimental): CBT101 cells, every 2 weeks
  Interventions: Biological: CBT101 cells, every 2 weeks
- CBT101 q4w (Experimental): CBT101 cells, every 4 weeks
  Interventions: Biological: CBT101 cells, every 4 weeks

INTERVENTIONS:
Biological: CBT101 cells, every 2 weeks — CBT101 cells, every 4 weeks
  Arms: CBT101 q2w
Biological: CBT101 cells, every 4 weeks — CBT101 cells, every 4 weeks
  Arms: CBT101 q4w

SUMMARY:
The objective of the study is to evaluate tolerability and safety of CBT101 in patients who underwent curative surgery and adjuvant therapy for solid cancer

ELIGIBILITY:
Inclusion Criteria:

1. Male and female adults aged 19 years and older
2. Patients with solid tumors as below (1) histologically or cytologically confirmed solid tumors (2) 4 - 12 weeks of last adjuvant therapy after radical operations and adjuvant therapy
3. Life expectancy 6 months
4. Eastern Cooperative Oncology Group perfornace status (ECOG PS) 0-1

Exclusion Criteria:

1. History of leptomeningeal carcinomatosis or spinal cord compression
2. History of peritoneal carninomatosis
3. Hemoglobine less than 9.0g/dL
4. Absolute Neutrophil Count (ANC) less than 1.5x10^3/mm^3
5. Platelet count less than 75x10^9/L
6. Total bilitbinn grater than 1.5 times te upper limit of normal
7. Alanine amino transferase (ALT) greater than 3 times the upper limit of normal
8. Alanine phospatase (ALP) greater than 2.5 times the upper limit of normal
9. Uncontrolled hypertension
10. Intensive insuline therapy
11. Active infectious disease
12. Patients with hypersensitivity history or allergy to investigational product
13. Pregmant of lactating woman
14. Patients who have participated in another clinical trials witin 30 days before the start of this clinical trial
15. Patients judged to be inappropriate for this study by the investigator with other reasons

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2020-09-21 (Actual); Primary Completion 2021-10-26 (Actual); Study Completion 2021-10-26 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) | 29 days
  Dose limiting toxicity (DLT)

SECONDARY OUTCOMES:
Disease-free survival rate (DFS) | 6 months
  Disease-free survival rate (DFS)
Oerall survival rate (OS) | 6 months
  Oerall survival rate (OS)

CONTACTS AND LOCATIONS:
Overall Officials: Chan Kim, Principal Investigator — CHA Bundang Medical Center
Locations (1):
- CHA Bundang Medical Center, Seongnam-si, Gyeonggi-do, South Korea